CLINICAL TRIAL: NCT02993081
Title: REFRACTIVE CHANGES AFTER CAPSULOTOMY WITH YAG LASER
Brief Title: Capsulotomy YAG Laser
Acronym: RCYAG
Status: Completed | Type: Observational
Sponsor: Instituto de Olhos de Goiania (Other)
Responsible Party: Sponsor
Other Study IDs: ARVO R1 2017
Record Dates: First submitted 2016-12-12; First posted 2016-12-15 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Refractive and Accommodative Disorders
Keywords: YAG laser

SUMMARY:
Study of refractive changes after capsulotomy with YAG laser in facectomized patients.

DETAILED DESCRIPTION:
A retrospective, quantitative study was carried out by analyzing the medical records of a reference ophthalmologic hospital in Goiás. Data from the pre and post YAG laser refractive index data were collected from 67 eyes of 66 patients analyzed in the period from May to November 2016.

We studied 67 eyes of 66 patients , both men and women , and 32 ( 47,7%) underwent myopia after the capsulotomy procedure with YAG laser and 25 ( 37.3%) hypermetropization and 10 (14.9%) maintained the refraction. The difference in refraction was found by the arithmetic mean of the spherical equivalent for the precapsulotomy procedure of -28.85D and post-capsulotomy of -31.75 D , giving a difference of -2.9 .

It was concluded with this study that the use of posterior capsulotomy with YAG laser post facectomy caused changes in the refraction of the patients studied, presenting myopia with greater frequency in the results. With these data, we observed the need for other future studies with a large number of eyes to prove what happened in this study.

ELIGIBILITY:
Inclusion Criteria: Complete data information about refraction and the date of the YAG laser -

Exclusion Criteria: Incomplete data

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We studied 67 eyes of 66 patients , both men and women by analyzing the medical records of a reference ophthalmologic hospital in Goiás.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2016-05; Primary Completion 2016-05 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Refractive changes after capsulotomy with YAG laser | 6 months